CLINICAL TRIAL: NCT01671540
Title: Evaluation of the Effects of Intrapulmonary Percussive Ventilation Using Functional Respiratory Imaging
Brief Title: Effects of IPV Assessed With Functional Imaging
Acronym: IPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Artesis University College, Antwerp (Other); FLUIDDA nv (Industry)
Responsible Party: Principal Investigator, Wilfried De Backer, Prof. Dr., University Hospital, Antwerp
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PML_Kine_IPV; artesis_G018 (Other: artesis university college)
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; IPV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrapulmonary percussive ventilation (Experimental): IPV is applied for 1 week (once a day) during the physical therapy treatment of the patient
  Interventions: Device: intrapulmonary percussive ventilation
- standard airwy claerance regime (Active Comparator): The standard treatment consists out of existing drainage techniques to remove secretion out of the lungs by means of breathing control exercises
  Interventions: Other: standard treatment

INTERVENTIONS:
Device: intrapulmonary percussive ventilation
  Other Names: IMP 2 by Breas Sweden
  Arms: Intrapulmonary percussive ventilation
Other: standard treatment — breathing control exercises
  Other Names: Autogenic drainge
  Arms: standard airwy claerance regime

SUMMARY:
In this study the invetigators seek an answer on the following hypothesis:

* What are the long term effects of an IPV treatment evaluated with classical outcome parameters? (FEV1, Raw)
* Is the possible effect noticeable on the novel technique and is this comparable with the classical outcome parameters?

DETAILED DESCRIPTION:
A Multicenter study conducted in university Hospital Antwerp (UZA) and ZNA Middelheim.

Tests are taken before and after one week IPV treatment. IPV is applied for 1 week during the physical therapy treatment of chronic obstructive pulmonary desease (COPD) patients admitted to the hospital for an excarebation. The IPV treatment is an additional treatment upon the standard treatment of the patients. The standard treatment consists out of existing drainage techniques to remove secretion out of the lungs by means of breathing control exercises. Patients are randomized into either the experimental group or the control group. The control group receives a standard physical therapy treatment without additional IPV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the hospital for a acute exacerbation
* Mild to severe COPD

Exclusion Criteria:

* Ischemic / ventricular aritmic
* Tracheotomise
* Pneumothorax
* Facial deformity
* Recent nose, mouth or ear operations
* Recent gastric operations.
* Intubated
* Epilepsy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Lung function testing | baseline and after one week
  (spirometric , bodybox en diffusion) Performed in the lung function laboratory according to ERS standards using Jaeger 5.1 device vital capacity (VC), FEV1, FEV1/VC, peak expiratory flow (PEF), MMEF 75/25, MEF 50, MEF 25, MIF 50, RV, total lung capacity (TLC), functionale residual capacity (FRC), resistance, spec resistance, TCO, alveolar volume (VA), TCO/VA, Maximal inspiratory pressure, Maximal expiratory pressure

SECONDARY OUTCOMES:
functional respiratory imaging | at baseline and after one week
  A 3D CT-scan is take. Images are uploaded into a software program for post processing 3D images are made and images are post processed

OTHER OUTCOMES:
questionnaires | 1 week
  St george Borg MRC

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, Phd, Principal Investigator — UZA pneumology
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium